CLINICAL TRIAL: NCT05582343
Title: Modified Interactive Screening Program Plus MINDBODYSTRONG: A Mental Health Resiliency Intervention for Nurses
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: American Foundation for Suicide Prevention (Other); University of San Diego (Other)
Responsible Party: Principal Investigator, Bernadette Melnyk, Dean and Helene Fuld Health Trust Professor of Evidence-Based Practice, College of Nursing Professor of Pediatrics & Psychiatry, College of Medicine Executive Director, the Helene Fuld Health Trust National Institute for EBP, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021B0417; TBT-2-007-21 (Other Grant/Funding Number: American Foundation for Suicide Prevention)
Record Dates: First submitted 2022-10-13; First posted 2022-10-17 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Suicide Threat; Burnout, Professional; Depression
Keywords: nurse; suicide; depression; burnout; trauma; computerized; CBT; intervention; depression screening
MeSH Terms: conditions — Burnout, Professional; Depression; Suicide; Burnout, Psychological; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Longitudinal, randomized RCT with repeated measures
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mISP (No Intervention): Participants who are identified as having moderate to high risk of suicide, as identified by suicide risk on the ISP, will be contacted by a mental health counselor who will engage them through the mISP encrypted interface online. The mental health counselor will offer counseling online through encryption or on the phone. Where indicated, the mental health counselor will provide the crisis hotline, and encourage participants to use their insurance provider and/or Employee Assistance Program to obtain treatment. The mental health counselor will offer to help with referrals and will bridge high-risk participants into treatment. Participants who are not identified as having moderate to high risk of suicide will be thanked for their time.
- mISP plus MINDSTRONG (Active Comparator): Participants identified as having a moderate to high risk of suicide based on ISP screening will then be randomized. Participants randomized to the MINDBODYSTRONG© program (intervention) will receive the 8-session online interactive program. Reminders will be sent weekly to complete the next MINDBODYSTRONG© session and a MINDBODYSTRONG© trained coach will check in with participants by phone at baseline, weeks 3 and 5 of the on-line program to reinforce key program concepts and assess whether participants are completing the weekly skills building activities. Nurses assigned to the control group will only receive the mISP alone (aforementioned) and will be contacted for follow-up surveys.
  Interventions: Behavioral: MINDBODYSTRONG™

INTERVENTIONS:
Behavioral: MINDBODYSTRONG™ — Digitalized MINDBODYSTRONG™ is designed for self-paced weekly use via an online platform.
  MINDBODYSTRONG© Session Content
  1. Thinking, feeling, & behaving, The ABCs of CBT, Mindfulness Skills Building: Positive self-talk/The ABCs
  2. Self-esteem & positive self-talk, Intentional gratitude, Managing change Skills building: Self-esteem & positive self-talk
  3. Stress, Healthy coping, Abdominal breathing Skills Building: Managing stress
  4. Problem solving, Setting goals, Steps to problem solving Skills building: Strategies to overcoming barriers
  5. Dealing w/ emotions in healthy ways, Using guided imagery, Coping strategies, Effective communication Skills building: Dealing with emotions
  6. Coping w/ stressful situations/valuable sleep Skills building: Coping w/ stressful situations
  7. Distress tolerance & added emotional regulation skills Skills bulding: RAIN practice, Self-love skill, Distracting using ACCEPTS
  8. Putting it all together for a healthy YOU!
  Other Names: COPE
  Arms: mISP plus MINDSTRONG

SUMMARY:
The overall purpose of this study is to evaluate the efficacy of an intervention designed to prevent nurse suicide. This randomized controlled trial will test the modified Interactive Screening Program (mISP) alone and the mISP combined with a program called MINDBODYSTRONG.

The mISP is a method of screening to detect clinicians at moderate to high risk for suicide and referring them for treatment through an encrypted anonymous on-line platform. MINDBODYSTRONG© is an adaptation of a well-tested cognitive-behavioral skills building intervention (also known as COPE in the literature) that provides a cognitive-behavior theory-based approach to decrease depression, anxiety and suicidal ideation and improve healthy lifestyle beliefs and behaviors in at-risk populations. MINDBODYSTRONG© will involve eight self-paced computerized sessions designed specifically for nurses and clinicians. Nurses will be recruited nationally through the professional nursing organizations and health systems.

DETAILED DESCRIPTION:
The study will be the first to test the combination of the mISP with a new on-line digitalized version of the previously tested manualized version of the CBSB program (i.e., MINDBODYSTRONG©) for nurses. If found to be effective, the combined program will be able to be easily scaled to prevent suicide in nurses and potentially other high-risk populations of clinicians. Although CBT is gold standard evidence-based treatment for depression, only a small percentage of affected individuals receive it due to a shortage of mental health providers, which contributes to high depression relapse rates of 50 to 70%. A scalable digitalized intervention could be one key solution to bringing CBT skills to nurses at risk for suicide who could so benefit from them. This randomized controlled trial (RCT) will determine the effects of the mISP, this adaptation of the American Foundation for Suicide Prevention's (AFSP) Interactive Screening program (ISP), combined with the on-line version of the MINDBODYSTRONG© program versus the HEAR program alone on depression, suicidal ideation, burnout, anxiety, post-traumatic stress, healthy lifestyle beliefs, healthy lifestyle behaviors, and job satisfaction in U.S. nurses.

ELIGIBILITY:
Inclusion Criteria:

* self-identify as a registered nurse
* identified as moderate to high risk of suicide by the mISP-specific interactive screening program assignment

Exclusion Criteria:

* low risk of suicide by the mISP-specific interactive screening program assignment
* under the age of 18 years
* prior participation in MINDBODYSTRONG
* prior participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 849 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change is being assessed for an increase or decrease in self-reported suicidal intent | Baseline (Timepoint 0), 8 weeks after baseline (Timepoint 1), 3 months after screening (Timepoint 2), 6 months after screening (Timepoint 3), 12 months after screening (Timepoint 4)
  The valid and reliable Columbia Suicide Severity Rating Scale assesses the severity of suicidal ideation and behavior through a semi-structured list of yes or no questions divided into four constructs: (1) suicidal ideation; (2) intensity of ideation; (3) suicidal behavior; and (4) suicidal lethality subscale (actual or potential).
Change in is being assessed for an increase or decrease in self-reported depressive symptoms | Baseline (Timepoint 0), 8 weeks after baseline (Timepoint 1), 3 months after screening (Timepoint 2), 6 months after screening (Timepoint 3), 12 months after screening (Timepoint 4)
  The 9-item valid and reliable Personal Health Questionnaire-9 will be used to measure depressive symptoms. Participants are asked to respond to nine items (e.g., little interest or pleasure in doing things; feeling down, depressed or hopeless) regarding how they have felt over the previous 2-week period. Scores are based on a 4-point Likert scale ranging from 0 "not at all" to 3 "nearly every day."

SECONDARY OUTCOMES:
Change in being assessed for an increase or decrease in self-reported anxiety symptoms | Baseline (Timepoint 0), 8 weeks after baseline (Timepoint 1), 3 months after screening (Timepoint 2), 6 months after screening (Timepoint 3), 12 months after screening (Timepoint 4)
  The valid and reliable Generalized Anxiety Disorder Scale (GAD-7) will be used to measure anxiety. The GAD-7 measures feelings and actions associated with anxiety within the prior 2-week period. Responses are based on a 4-point Likert scale ranging from 0 (not at all) to 3 (nearly everyday).
Change is being assessed for an increase or decrease in self-reported burnout level | Baseline (Timepoint 0), 8 weeks after baseline (Timepoint 1), 3 months after screening (Timepoint 2), 6 months after screening (Timepoint 3), 12 months after screening (Timepoint 4)
  The following non-proprietary single-item question from the Maslach Burnout Inventory will be used to measure burnout: "Overall, based on your definition of burnout, how would you rate your level of burnout?" Responses are scored on a five-category ordinal scale, where 1 = "I enjoy my work. I have no symptoms of burnout;" 2 = "Occasionally I am under stress, and I don't always have as much energy as I once did, but I don't feel burned out;" 3 = "I am definitely burning out and have one or more symptoms of burnout, such as physical and emotional exhaustion;" 4 = "The symptoms of burnout that I'm experiencing won't go away. I think about frustration at work a lot;" and 5 = "I feel completely burned out and often wonder if I can go on. I am at the point where I may need some changes or may need to seek some sort of help."
Change is being assessed for an increase or decrease in self-reported post-traumatic stress levels | Baseline (Timepoint 0), 8 weeks after baseline (Timepoint 1), 3 months after screening (Timepoint 2), 6 months after screening (Timepoint 3), 12 months after screening (Timepoint 4)
  The Primary Care PTSD Screen for DSM-5 (PC-PTSD-5) will be used to screening for post-trauma symptoms. This 5-item screening tool was developed to identify individuals with probable PTSD in a primary care setting.
Change is being assessed for an increase or decrease in self-reported job satisfaction | Baseline (Timepoint 0), 8 weeks after baseline (Timepoint 1), 3 months after screening (Timepoint 2), 6 months after screening (Timepoint 3), 12 months after screening (Timepoint 4)
  Job Satisfaction will be measured using the Job Satisfaction Scale (JSS). This 7-item scale queries responses such as "I find real enjoyment in my job" and are measured on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree).
Change is being assessed for an increase or decrease in self-reported healthy lifestyle beliefs | Baseline (Timepoint 0), 8 weeks after baseline (Timepoint 1), 3 months after screening (Timepoint 2), 6 months after screening (Timepoint 3), 12 months after screening (Timepoint 4)
  The Healthy Lifestyle Beliefs Scale is a 10-item scale that will be used to tap cognitive beliefs about dealing with stress/problems and engaging in healthy lifestyle behaviors, the proposed mediator in this study. Participants respond to each of the items on a 10-point Likert scale ranging from (1) strongly disagree to (5) strongly agree.
Change is being assessed for an increase or decrease in self-reported healthy lifestyle behaviors | Baseline (Timepoint 0), 8 weeks after baseline (Timepoint 1), 3 months after screening (Timepoint 2), 6 months after screening (Timepoint 3), 12 months after screening (Timepoint 4)
  The Healthy Lifestyle Behaviors scale is a 16-item scale that asks for responses on statements such as "I make healthy food choices" and "I set goals I can accomplish." It us scored on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree).
Open-ended stressors question | Baseline (Timepoint 0), 8 weeks after baseline (Timepoint 1), 3 months after screening (Timepoint 2), 6 months after screening (Timepoint 3), 12 months after screening (Timepoint 4)
  One previously tested question on self-reported stressors (risk factors) will be used. The question is: Please take a minute to let us know about anything that has been particularly stressful for you lately - death of a loved one, relationship break-up, academic stressors, family or money problems, difficulty with your living situation - or anything else that might be contributing to how you are feeling.
Evaluation Questionnaire | 3 months after screening (Timepoint 2), 6 months after screening (Timepoint 3), 12 months after screening (Timepoint 4)
  . A questionnaire also will be administered to yield open ended feedback on the interventions in terms of their helpfulness as well as collect data on whether the nurses have received any treatment since beginning the study (e.g., therapy, medication).

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Melnyk BM, Davidson JE, Mayfield C, Zisook S, Tucker S, Hsieh AP, Cooper A, Gray-Bauer R, Hoying J, Cuccia AF, Tan A. A study protocol for the modified interactive screening program plus MINDBODYSTRONG(c) RCT: A mental health resiliency intervention for nurses. PLoS One. 2024 Jun 6;19(6):e0303425. doi: 10.1371/journal.pone.0303425. eCollection 2024. PMID 38843149